CLINICAL TRIAL: NCT02025296
Title: Ubiquitous Healthcare Service With Multifactorial Intervention in Diabetes Care: a Randomized Controlled Trial
Brief Title: Ubiquitous Healthcare Service With Multifactorial Intervention in Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U-healthcare system
Record Dates: First submitted 2013-12-23; First posted 2014-01-01 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus With Hypoglycemia
Keywords: Telemedicine; Clinical decision support system; Ubiquitous healthcare; Diabetes Care; Multifactorial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Monitoring of Blood Glucose (No Intervention): measurement of their blood glucose level using a glucometer at least eight times a week
- U-healthcare (Experimental): individualized multidisciplinary u-healthcare service combined with exercise monitoring and dietary feedback on glucose control
  Interventions: Device: U-healthcare

INTERVENTIONS:
Device: U-healthcare — use of a public switched telephone network (PSTN)-connected glucometer to measure their blood glucose level at the same frequency as the SMBG group
  Arms: U-healthcare

SUMMARY:
Recently, we generated a new multidisciplinary ubiquitous healthcare system by upgrading our clinical decision supporting system (CDSS) rule engine, and integrating a physical activity-monitoring device and dietary feedback into a comprehensive package. We hypothesize that individualized multidisciplinary u-healthcare service combined with exercise monitoring and dietary feedback will result in better glucose control with less hypoglycemia in an elderly population.

DETAILED DESCRIPTION:
The use of telemedicine (also known as connected health, e-health, or telehealth) has been proven to be beneficial in chronic disease management. Now, the classic concept of telemedicine has been evolving to ubiquitous (u)-healthcare system with advanced information technologies which provides real-time individualized feedback using a monitoring device attached to the internet or a mobile phone system.

A few studies showed that adopting a u-healthcare system helped patients improve their blood glucose control and reduced hypoglycemia or weight gain. In a previous study, supervised telemonitoring was effective for blood pressure control in hypertensive patients in primary care settings. A recent study showed that telemonitoring with pharmacist's help achieved better blood pressure control compared with usual care during 12 months of intervention.

A clinical decision support system (CDSS) is the key to this system, building up an individualized CDSS rule engine is the crux of the u-healthcare system because current glucose control status, antidiabetic medications, lifestyle, and severity of hypoglycemia vary between individual patients.

Recently, our u-healthcare team generated a new multidisciplinary u-healthcare system by upgrading the CDSS rule engine, and integrating a physical activity-monitoring device and dietary feedback into a comprehensive package. With this integrated system, we investigate the effect of individualized multidisciplinary u-healthcare service combined with exercise monitoring and dietary feedback on glucose control with less hypoglycemia in Korean elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus
* Glycated hemoglobin (HbA1c) levels: 7.0-10.5%

Exclusion Criteria:

* Patients who were unable to use text messages or to access the internet for any reason

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
proportion of patients achieving the target of HbA1c <7% without hypoglycemia | 6 months
  The primary endpoint of the present study was the proportion of patients achieving the target of HbA1c <7% without hypoglycemia at 6 months.

SECONDARY OUTCOMES:
Hypoglycemia | 6 months
  Numbers of hypoglycemic events
Obesity index | 6 months
  Changes of BMI and Waist circumference
Lifestyle | 6 months
  Changes of caloric intake and exercise

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, PhD, Principal Investigator — SNUBH
Locations (1):
- SNUBH, Seongnam-si, Gyeonggi-do, South Korea